CLINICAL TRIAL: NCT07222358
Title: Multi-component Remote Assessment in Adult Survivors Using a Connected Technology Platform for Healthcare Delivery
Status: Not yet recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RAIS
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Childhood Cancer
Keywords: St. Jude Alumni; St. Jude Life Participants
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A one-time blood sample (30 mL) will be collected from each participant either at home or at a local facility. The sample will include clinical laboratory tests such as Complete Blood Count (CBC), Comprehensive Metabolic Panel (CMP), lipids, HbA1c, and N-terminal pro-B-type natriuretic peptide (NT-proBNP). The remaining portion of the sample will be banked at St. Jude Children's Research Hospital for future research.
  Retained blood samples may contain DNA and could be used for future genetic or molecular analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remote Monitoring Group: Participants will undergo a 12-week remote monitoring program using wearable devices and complete surveys and a one-time lab draw. A subset will participate in interviews post-intervention.
  Interventions: Behavioral: Remote Monitoring Program

INTERVENTIONS:
Behavioral: Remote Monitoring Program — * Participants receive devices (Apple Watch, blood pressure monitor, Continuous Glucose Monitor (CGM), scale, measuring tape).
  * Monitoring includes ECG, blood pressure, glucose, weight, waist circumference, physical activity, and sleep.
  * Surveys include health status, medication use, personality traits, and acceptability measures.
  * One-time blood draw includes CBC, CMP, lipids, HbA1c, NT-proBNP
  * Food logging during CGM use.
  * Semi-structured interviews post-study for a subset.

SUMMARY:
This feasibility study evaluates a 12-week, multi-component remote assessment program for adult survivors of childhood cancer. The study aims to determine the participation and adherence rates to remote monitoring of cardiometabolic health using wearable devices, surveys, and laboratory testing facilitated by a third-party vendor.

Primary Objective - To establish the feasibility of a multi-component remote assessment program for adult survivors.

* The primary outcome for feasibility will be the participation rate (# eligible survivors approached who enroll) and completion rate (# of eligible survivors who enroll and remain on study through completion).
* An additional outcome for feasibility will be adherence to the multicomponent remote assessment among participants.

Secondary Objective

* To estimate the proportion of participants who complete each individual study component (adherence to each individual component monitoring).

DETAILED DESCRIPTION:
Survivors of childhood cancer face increased risks of late effects, including cardiometabolic conditions. Due to geographic diversity and mobility limitations, remote research participation is essential. This study pilots a remote assessment platform to monitor cardiometabolic health indicators such as blood pressure, heart rate variability, glucose control, physical activity, sleep, diet, and laboratory biomarkers. Participants will be on-boarded by a vendor, receive devices, and complete assessments remotely. A subset will participate in interviews to evaluate platform acceptability and barriers. The study will assess feasibility through participation and adherence rates, aiming to inform future remote intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥18 years of age
* Participant is enrolled in the St. Jude Life (SJLIFE) cohort
* Participant is able and willing to provide informed consent
* Participant has signed a separate consent for the St. Jude banking protocol (TBANK)
* Participant received anthracycline (≥100 mg/m²), chest or abdominal radiation as part of childhood cancer treatment
* Participant owns a SmartPhone compatible with the vendor platform, Apple HealthKit, and Dexcom (a wearable device that continuously tracks glucose levels)
* Participant verbalizes understanding directions for completing remote study activities with the third-party partner
* Participant is fluent in English

Exclusion Criteria:

* Participant uses a continuous glucose monitor for diabetes management or has diabetes requiring insulin or more than 1 agent for treatment at baseline
* Participant is currently enrolled on an intervention or active longitudinal monitoring ancillary study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Participation rate | Assessed at contact for enrollment of each participant (baseline/screening).
  The proportion of eligible survivors approached who enroll in the intervention
On-boarding rate | Baseline at study entry through week 12
  The proportion of consented participants who successful onboard with the vendor and contribute any study data beyond baseline
Completion rate | Baseline at study entry through week 12
  The proportion of enrolled survivors who remain on study and complete both baseline and week 12/end of study assessments.
Adherence to the remote monitoring intervention | Baseline at study entry through week 12
  The proportion of enrolled survivors who complete at least 2/3 of the pre-specified remote monitoring study components

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Dixon, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols